CLINICAL TRIAL: NCT04252885
Title: A Randomized, Open-label, Controlled Study of the Efficacy of Lopinavir Plus Ritonavir and Arbidol for Treating With Patients With Novel Coronavirus Infection
Brief Title: The Efficacy of Lopinavir Plus Ritonavir and Arbidol Against Novel Coronavirus Infection
Acronym: ELACOI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou 8th People's Hospital (Other)
Responsible Party: Principal Investigator, Linghua LI, Vice chief of Infectious Disease Center, Guangzhou 8th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GZ8H-V1.0 20200122
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Coronavirus Infections
Keywords: Coronavirus infection; Lopinarvir plus ritonavir; Arbidol; Efficacy
MeSH Terms: conditions — Coronavirus Infections | interventions — Lopinavir; Ritonavir; umifenovir

STUDY DESIGN:
Intervention Model Description: 125 patients are randomized in 3 groups (2:2:1). In group A(Standard treatment+lopinavir/ritonavir) , 50 cases are given ordinary treatment plus a regimen of lopinavir (200mg) and ritonavir (50mg) (oral, q12h, every time 2 tablets of each, taking for 7-14 days). In group B (Standard treatment+arbidol), 50 cases are given ordinary treatment plus a regimen of arbidol (100mg) (oral, tid, 200mg each time, taking for 7-14 days). In group C (Standard treatment）, 25 cases are only given ordinary treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A-Standard treatment+lopinavir/ritonavir (Experimental): In group A, 50 cases are given ordinary treatment plus a regimen of lopinavir (200mg) and ritonavir (50mg) (oral, q12h, every time 2 tablets of each, taking for 7-14 days).
  Interventions: Drug: Lopinavir and Ritonavir Tablets
- Group B-Standard treatment+arbidol (Active Comparator): In group B, 50 cases are given ordinary treatment plus a regimen of arbidol (100mg) (oral, tid, 200mg each time, taking for 7-14 days).
  Interventions: Drug: Arbidol
- Group C-Standard treatment (No Intervention): In group C, 25 cases are only given ordinary treatment.

INTERVENTIONS:
Drug: Lopinavir and Ritonavir Tablets — As indicated in arm/group descriptions
  Other Names: Kletra
  Arms: Group A-Standard treatment+lopinavir/ritonavir
Drug: Arbidol — As indicated in arm/group descriptions
  Arms: Group B-Standard treatment+arbidol

SUMMARY:
The study explores the efficacy of lopinavir plus ritonavir and arbidol in treating with novel coronavirus infection. As a result this study would provide evidence for the clinical usage of these drugs in the future .

DETAILED DESCRIPTION:
This is a phase IV, open-labelled, randomized controlled clinical trial. A total of 125 cases who are novel coronavirus positive are planned to be recruited. These cases are randomized into 3 groups: in group A（Standard treatment+lopinavir/ritonavir）, 50 cases are given ordinary treatment plus a regimen of lopinavir (200mg) and ritonavir (50mg) (oral, q12h, every time 2 tablets of each, taking for 7-14 days). In group B（Standard treatment+arbidol） , 50 cases are given ordinary treatment plus a regimen of arbidol (100mg) (oral, tid, 200mg each time, taking for 7-14 days). In group C（Standard treatment）, 25 cases are only given ordinary treatment. The observation duration is 21 days. Patients will be followed up at baseline (day 0) and day 2, 4, 7, 10,14, 21 after receiving indicated treatment. The primary observed indicators include viral nucleic in acid nose / throat swab, body temperature, respiratory rate, oxygen saturation of blood, chest imaging. The secondary observed indicators include but not limited to blood pressure, heart rate, blood routine test, liver and kidney function, myocardial enzyme, flow cytometry classification and counting, cytokines, other infection indicators, conditions and parameters of auxiliary respiration, the total days in hospital, exacerbation and mortality.

ELIGIBILITY:
Inclusion Criteria:

* In sputum, throat swab, lower respiratory tract secretion, blood and other samples, the nucleic acid of the novel coronavirus was positive, or the sequencing of the virus gene was highly homologous with the known novel coronavirus
* Age is between 18-80 years old, the weight is more than 30kg, and there is no limit for men and women
* The following conditions were met: creatinine ≤ 110 umol / L, creatinine clearance rate (EGFR) ≥ 60 ml / min / 1.73m2, AST and ALT ≤ 5 × ULN, TBIL ≤ 2 × ULN;
* The subjects should fully understand the purpose, nature, method and possible reaction of the study, voluntarily participate in the study and sign the informed consent.

Exclusion Criteria:

* Have a clear history of lopinavir or ritonavir or arbidol allergy
* Severe nausea, vomiting, diarrhea and other clinical manifestations affect the oral or absorption of the drugs
* At the same time, take drugs that may interact with lopinavir or ritonavir or arbidol
* Patients with serious underlying diseases, including but not limited to heart disease (including history of angina pectoris or coronary heart disease or myocardial infarction, atrioventricular block), lung, kidney, liver malfunction and mental diseases that cannot be treated together
* ancreatitis or hemophilia
* Pregnant and lactating women
* Suspected or confirmed history of alcohol and drug abuse
* Participated in other drug trials in the past month
* The researchers judged that patients were not suitable for the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
The rate of virus inhibition | Day 0, 2, 4, 7, 10, 14 and 21
  Novel coronaviral nucleic acid is measured in nose / throat swab at each time point.

SECONDARY OUTCOMES:
The disease prorogation-temperature | Day 0 till day 21
  Body temperature will be followed everyday during time frame.
The disease prorogation-respiratory function 1 | Day 0 till day 21
  Respiratory rate will be followed everyday during time frame.
The disease prorogation-respiratory function 2 | Day 0 till day 21
  Oxygen saturation of blood will be followed everyday during time frame.
The disease prorogation-respiratory function 3 | Day 0, 4, 7, 10, 14 and 21
  Chest imaging will be taken at each time point.

OTHER OUTCOMES:
Patients health condition-routine test | Day 0 till day 21
  Blood pressure and heart rate will be followed everyday during time frame.
Patients health condition-liver function | Day 0, 4, 7, 10, 14 and 21
  Liver function will be assessed as AST, ALT and TBIL at each time point.
Patients health condition-kidney function | Day 0, 4, 7, 10, 14 and 21
  Kidney function will be assessed as eGFR and creatine clearance rate at each time point.
Patients health condition-other blood routine test | Day 0, 4, 7, 10, 14 and 21
  Blood routine and myocardial enzyme will be measured at each time point.
Patients health condition-blood routine test | Day 0, 4, 7, 10, 14 and 21
  Flow cytometry classification and counting and cytokines will be measured at each time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Eighth People's Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Li Y, Xie Z, Lin W, Cai W, Wen C, Guan Y, Mo X, Wang J, Wang Y, Peng P, Chen X, Hong W, Xiao G, Liu J, Zhang L, Hu F, Li F, Zhang F, Deng X, Li L. Efficacy and Safety of Lopinavir/Ritonavir or Arbidol in Adult Patients with Mild/Moderate COVID-19: An Exploratory Randomized Controlled Trial. Med. 2020 Dec 18;1(1):105-113.e4. doi: 10.1016/j.medj.2020.04.001. Epub 2020 May 19. PMID 32838353